CLINICAL TRIAL: NCT02564159
Title: Ultrasound Measurement of the Quadriceps Muscle Diameter for the Detection and the Follow-up of Malnutrition in Patients Receiving Mechanical Ventilation in Intensive Care Unit
Brief Title: Malnutrition Screening by Muscle Ultrasound in Patients Requiring Mechanical Ventilation in Intensive Care Unit
Acronym: MALICUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC14_0424
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Malnutrition; Critical Illness
Keywords: malnutrition; muscle ultrasound; intensive care unit; mechanical ventilation; albumin; prealbumin; nutrition
MeSH Terms: conditions — Malnutrition; Critical Illness | interventions — High-Energy Shock Waves; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-risk patient for malnutrition acquired in ICU (Experimental): Patients admitted in ICU and treated with mechanical ventilation with expected duration of 48 hours or more
  Interventions: Other: Measure of quadriceps thickness with ultrasonography and albumin/prealbumin levels
- Controls patients: Elective surgery (Other): Controls patients: Elective surgery (neurosurgery, thoracic surgery, vascular surgery)
  - Patients admitted in a post-operative care unit of the university hospital of Nantes after elective surgery with expected duration ICU length of stay < 48 hours
  Interventions: Other: Measure of quadriceps thickness with ultrasonography and albumin/prealbumin levels

INTERVENTIONS:
Other: Measure of quadriceps thickness with ultrasonography and albumin/prealbumin levels — * Evaluation of quadriceps diameter on the anterior aspect of the thigh using the mid-distance between the anterior superior iliac spine and the upper pole of the patella ;
  * Biospecimen collection: Blood samples (prealbumin levels, C-reactive protein, Interleukin-1, Interleukin-6, TNF-alpha and PATROL test™)collection of albumin and prealbumin levels

SUMMARY:
Malnutrition is a major risk factor for morbidity and mortality of patients managed in intensive care unit. Early recognition and treatment of adult malnutrition are recommended in acute care settings especially for patients requiring mechanical ventilation. Biochemical indicators like serum concentrations of albumin and prealbumin (transthyretin) have a tradition of being used as markers of nutritional status but remains influenced by nonnutritional factors. A recent assessment of quadriceps muscle diameter with ultrasound method has gained interest for screening and follow-up of muscle weakness at the bedside in critically ill patients. In this light, the MALICUS project aims to investigate the validity of ultrasound as measurement tool for assessing malnutrition acquired in intensive care unit.

Skeletal muscle is central to cytokine regulation and it contributes 85% of total body glucose clearance. Some research findings suggest that muscle wasting is a smoldering inflammatory state partially driven by cytokines and oxidative stress but these conclusions need to be investigated in context of critically ill patients and perioperative settings.

The investigators search to determine impact of inflammatory biomarkers (IL-1, IL-6 and TNF-α) and oxidative stress (evaluated by quantifying the global anti-oxidative defenses in patient with an original method (Patrol® test) based on the use of excited molecular oxygen (singlet oxygen) as a source of ROS on erosion of lean body mass measure with quadriceps muscle ultrasound. Consequently, in an ancillary study of the MALICUS project, the investigators wish to investigate interaction between acute inflammation and muscle wasting.

ELIGIBILITY:
Study Population

Subjects will be enrolled from 2 venues:

1. Adults ICU patients (> 18 years) requiring period of mechanical ventilation. Subjects affiliated with an appropriate social security system
2. Adults patients admit requiring ICU length of stay < 48h after eligible surgery

<!-- -->

1. MALICUS Study

   Inclusion Criteria:

   - Patient requiring invasive mechanical ventilation

   - Expected duration of ventilation longer than 48 hours

   - Age > 18 years
   * Subjects affiliated with an appropriate social security system

   Non inclusion Criteria:

   - Invasive mechanical ventilation started for more than 48 hours

   - Patient severely malnourished at baseline (at least one of the following criteria)
   * Prealbuminemia < 0,11 g/L
   * BMI ≤ 18,5 (or ≤ 22 beyond 70 years)
   * Unintentional weight loss > 5% in the previous month or > 10% in the last 6 months - Glomerular nephropathy history/nephrotic syndrome, chronic renal failure (MDRD < 30 ml/min), liver cirrhosis or exudative gastro-enteropathy - Glucocorticoid (> 10 mg / day of prednisone equivalent ) long-term therapy ( > 1 month) - Impossible ultrasound measure of anterolateral diameter for the two quadriceps muscles

     - Neuromuscular disease that can cause muscle atrophy at a lower limb, without any support in the ICU
2. Control group - BIOBANK-MALICUS

Inclusion criteria:

* Elective surgery requiring an ICU stay (neurosurgery, vascular surgery, thoracic surgery)
* Expected duration of ventilation shorter than 48 hours

Non inclusion criteria:

• Elective surgery with cardiopulmonary bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Sensitivity of ultrasound measurement of the quadriceps muscle anteroposterior diameter for the diagnosis of malnutrition in patients requiring mechanical ventilatory support in ICU | 8 days
  Anteroposterior diameter of the quadriceps muscle (mid-thigh distance between the anterior superior iliac spine and the upper pole of the patella) will be compared with biochemical method (prealbumin levels). Patients will be classified as true positive, true negative, false positive or false negative relative to the gold standard (biochemical method). The sensitivity and the specificity of ultrasound method to detect malnutrition will be calculated with their 95% confidence interval.

SECONDARY OUTCOMES:
Comparing measurement of quadriceps muscle diameter measure by ultrasound of the thigh and Interleukin 6 level | 8 days
  Biospecimen collection (serum) Blood serum for biological specimen of pro-inflammatory cytokines (IL-1, IL-6 and TNF-α), inflammatory proteins (C-Reactive Protein) and total oxidative stress (PATROL® test)
3. Comparing measurement of quadriceps muscle diameter measure by ultrasound of the thigh and NUTRIC-Score at baseline | 8 days
  NUTRIC-Score

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand ROZEC, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France